CLINICAL TRIAL: NCT01965327
Title: Open-label Pilot Study of Interferon Gamma-1b (Actimmune™) for the Treatment of Friedreich Ataxia (FRDA)
Brief Title: Interferon Gamma-1b in Friedreich Ataxia (FRDA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other); Vidara Therapeutics Research Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-010121; 13-010121 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2013-08-27; First posted 2013-10-18 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich ataxia; Interferon gamma-1b; FRDA
MeSH Terms: conditions — Friedreich Ataxia | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon Gamma-1b (ACTIMMUNE) (Experimental): All individuals in this study will be given active medication (interferon gamma-1b) for 12 weeks. This will be administered according to a dose-escalation schedule.
  Interventions: Drug: Interferon Gamma-1b

INTERVENTIONS:
Drug: Interferon Gamma-1b — Subjects will begin by taking 10 mcg/m2 of IFN-g-1b for the first two weeks of the study. Dose will be escalated to 25 mcg/m2 of IFN-g-1b for weeks three and four of the study. Finally, the dose will be escalated to 50 mcg/m2 of IFN-g-1b for the last eight weeks of the study, which is the current dose approved by the FDA for children.
  All doses will be administered via subcutaneous injection.
  Other Names: Actimmune™; IFN-g-1b

SUMMARY:
Friedreich ataxia (FRDA) is a progressive neurodegenerative disease of children and adults for which there is presently no therapy. Recently, a study reported that interferon gamma (IFN-g) could raise frataxin protein levels in both cell lines derived from patients with Friedreich ataxia and in a mouse model with Friedreich ataxia. The present study will test whether IFN-g is safe, tolerated and potentially efficacious in a heterogeneous cohort of children with FRDA.

DETAILED DESCRIPTION:
Study Objectives:

Primary:

• To assess the effect of Interferon Gamma-1b (IFN-g) on increasing frataxin expression and protein in children with FRDA.

Secondary:

* To assess the effect of IFN-g on neurological outcomes (FARS, performance measures, and hearing) in subjects with FRDA.
* To assess the effectiveness of IFN-g on quality of life in subjects with FRDA.
* To assess the safety and tolerability of IFN-g at the currently approved dose in the FRDA population.

Study Phases:

Screening - During screening, subjects will be assessed for inclusion and exclusion criteria.

Intervention - Subjects will begin treatment at baseline visit and the dose of study medication will be increased to the maximum dose over four weeks. The subjects will be maintained at the maximum dose for 8 weeks. After 12 weeks, treatment will stop. Study medication will be administered via subcutaneous injections three times per week for 12 weeks.

Follow-up - Follow-up visits will occur at 7 and 28 days after the subject has completed the 12 weeks of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with FRDA confirmed by genetic testing with 2 expanded Guanine-adenine-adenine repeats
* Females who are not pregnant or breast feeding, and who do not intend to become pregnant. Females of child-bearing potential must use a reliable method of contraception and must provide a negative urine pregnancy test at screening
* Stable doses of all medications, vitamins and supplements for 30 days prior to study entry and for the duration of the study
* Parent/guardian permission (informed consent) and child assent

Exclusion Criteria:

* Any unstable illness that in the investigator's opinion precludes participation in this study
* Use of any investigational product within 30 days prior to enrollment
* Subjects with a history of substance abuse
* Presence of clinically significant cardiac disease
* History of hypersensitivity to IFN-g or E. coli derived products
* Presence of severe renal disease or hepatic disease
* Clinically significant abnormal White blood cell count, hemoglobin or platelet count
* Any subject planning a scheduled surgical procedure during the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects were screened and all were enrolled in the study between September - December 2013.
Groups:
- Interferon Gamma-1b (ACTIMMUNE): All individuals in this study were treated with interferon gamma-1b (ACTIMMUNE). Doses were administered via subcutaneous injections three times per week for 12 weeks. Dose-escalation schedule was completed by all subjects as follows: For the first two weeks subjects took10 mcg/m2 of interferon gamma-1b (IFN-g-1b), then the dose was escalated to 25 mcg/m2 of IFN-g-1b for weeks three and four of the study, finally, the dose was escalated to 50 mcg/m2 of IFN-gamma-1b for the last eight weeks of the study, which is the current dose approved by the FDA for children.
Period: Overall Study
Arm/Group | Interferon Gamma-1b (ACTIMMUNE)
Started | 12
Completed | 10 (Prior to completion, 2 subjects were withdrawn by the PI for failure to adhere to study protocol.)
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Gamma-1b (ACTIMMUNE)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [8 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Blood Frataxin Levels
Description: Assessment of the change in whole blood frataxin levels as assessed by lateral flow assay using an immunoassay for frataxin. Frataxin levels in the blood were measured at each study visit. Change in frataxin level at the end of treatment (week 12) relative to frataxin level at baseline was analyzed.
Time Frame: Frataxin levels were measured at the beginning and conclusion of treatment (baseline and 12 weeks)
Population: The primary analysis was based on an intent-to-treat approach including all subjects who had baseline frataxin blood levels collected.
Measure: Mean (Standard Deviation); unit: percentage of baseline frataxin level
Arm/Group | Interferon Gamma-1b (ACTIMMUNE)
Number analyzed (Participants) | 12
percentage of baseline frataxin level | -1.5 (1.9)
Statistical Analysis 1: Comparison: Interferon Gamma-1b (ACTIMMUNE); Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Missing data were imputed by last observation carried forward

2. Secondary Outcome: Change in Total Friedreich Ataxia Rating Scale (FARS) Score
Description: The Friedreich Ataxia Rating Scale (FARS) is neurological rating scale specifically developed and validated for FRDA. The FARS includes assessments of stance, gait, upper and lower limb coordination, speech, proprioception and strength. In addition to the standard neurological examination, the FARS contains three quantitative performance measures and a component that assesses activities of daily living (ADL). Quantitative performance measures include the nine-hole peg test, and a timed 25-foot walk. FARS scores correlate significantly with functional disability, activities of daily living scores and disease duration. The scores from the three subscales are added to generate a total score ranging from 0 to 159, with a higher score indicating a greater level of disability.
Time Frame: FARS score was calculated at the beginning and conclusion of treatment (baseline and 12 weeks)
Population: The analysis was based on an intent-to-treat approach and included all subjects with baseline FARS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon Gamma-1b (ACTIMMUNE)
Number analyzed (Participants) | 12
units on a scale | -4.98 (3.6)
Statistical Analysis 1: Comparison: Interferon Gamma-1b (ACTIMMUNE); Test type: Superiority or Other; p = 0.0078, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: All subjects entered into the study (12) were included in the safety analysis. The frequencies of adverse events were summarized by type, body system, severity and relationship to study drug.
Arm/Group | Interferon Gamma-1b (ACTIMMUNE)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Gamma-1b (ACTIMMUNE) (N=12)
Absominal Pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Influenza like illness (Infections and infestations) | 6
Pyrexia (General disorders) | 2
Contusion (Skin and subcutaneous tissue disorders) | 1
Elevated transaminases (Investigations) | 1
Decreased Platelet Count (Blood and lymphatic system disorders) | 1
Decreased Appetite (General disorders) | 1
Myalgia (General disorders) | 4
Headache (General disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Injection Site Pain (Investigations) | 3
Injection Site Bruising (General disorders) | 4
Injection Site Dermititis (General disorders) | 1
Injection Site Discoloration (General disorders) | 1
Injection Site Edema (General disorders) | 1

LIMITATIONS AND CAVEATS:
This study was performed in a small population of children with Friedreich ataxia (n=12) and without a placebo arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes